CLINICAL TRIAL: NCT02582138
Title: Sarcopenia and Physical fRailty IN Older People: Multi-componenT Treatment Strategies (SPRINTT)
Brief Title: Multicomponent Intervention for Physical Frailty and Sarcopenia
Acronym: SPRINTT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Roberto Bernabei, Professor of Geriatrics, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 115621; IMI-JU-09-2013-02 (Other Grant/Funding Number: Innovative Medicine Initiative)
Record Dates: First submitted 2015-10-08; First posted 2015-10-21 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Sarcopenia
Keywords: physical frailty; sarcopenia; exercise; nutrition; information and communications technology
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multicomponent intervention (MCI) (Experimental): The multicomponent intervention will include a physical activity programme, a nutritional intervention and an information and communications intervention.
  Interventions: Other: Multicomponent intervention (MCI)
- Healthy Aging Lifestyle Education (HALE) (Active Comparator): The health aging lifestyle education programme will be based on workshops. Participants will receive information on a variety of topics of relevance to older persons (e.g., recommended preventive services and screenings at different ages). The programme will also include a short instructor-led programme (5-10 minutes) of upper extremity stretching exercises or some relaxation techniques that will be performed at the end of each workshop.
  Interventions: Other: Healthy Aging Lifestyle Education (HALE)

INTERVENTIONS:
Other: Multicomponent intervention (MCI) — The multicomponent intervention will include physical activity (PA), nutrition and information and communications technology (ICT). The PA will be of moderate intensity and will include aerobic, strength, flexibility, and balance training. Walking will be the primary mode of PA .
  The nutritional intervention will combine individual nutritional assessment and personalised dietary recommendations to achieve:
  * a daily total energy intake of 25-30 kcal/kg body weight;
  * an average protein daily intake between 1.0 and 1.2 g/Kg/body weight.
  The ICT component will involve the use of an ad hoc technological device to record actimetry data to support the elaboration of a personalised training programme.
  Arms: Multicomponent intervention (MCI)
Other: Healthy Aging Lifestyle Education (HALE) — The healthy aging lifestyle education programme will be based on a workshop series. Participants will receive information on a variety of topics of relevance to older adults (e.g., recommended preventive services and screenings at different ages). The programme will also include a short instructor-led programme (5-10 minutes) of upper extremity stretching exercises or some relaxation techniques that will be performed at the end of each workshop.
  Arms: Healthy Aging Lifestyle Education (HALE)

SUMMARY:
The SPRINTT study will evaluate the efficacy of a multicomponent intervention programme (physical activity, nutritional counselling/dietary intervention, and information and communications technology intervention) compared with a healthy aging lifestyle education programme on mobility disability, in non-disabled older people with physical frailty and sarcopenia.

DETAILED DESCRIPTION:
As the life expectancy in European countries continues to increase, the maintenance of physical independence in older persons has become a major public health priority. The ability to ambulate without assistance is crucial for independent living and it is often the first ability to be lost in the process leading to disability. Older people who have impaired walking function need more assistance and are more likely to be placed in nursing homes, have a higher risk of morbidity, mortality and hospitalisation, and experience a reduced quality of life. The ultimate goals of the Sarcopenia and Physical fRailty IN older people: multicomponenT Treatment strategies (SPRINTT) project are to offer efficient treatment options, based on a multicomponent intervention including physical activity, nutrition and information and communications technology, to physically frail, sarcopenic older persons and to improve their quality of life. The result will directly contribute to the long-term sustainability and efficiency of health- and social-care systems. The conceptualisation of physical frailty and sarcopenia (PF&S) as proposed in SPRINTT will promote significant advancements over the traditional approaches by enabling the precise operationalisation of the condition, a clear identification of the affected population and the rapid translation of findings to the clinical arena.

ELIGIBILITY:
Inclusion criteria:

1. Short Physical Performance Battery (SPPB) score between 3 (included) and 9 (included);
2. Able to complete the 400-m walk test within 15 min without sitting down, help from another person, use of a walker, or stopping for more than 1 minute at a time;
3. Presence of low muscle mass based on Dual Energy X-Ray Absorptiometry (DXA) scan, according to the Foundation for the National Institutes of Health Sarcopenia Project (FNIH) criteria:

   * Body mass index-adjusted appendicular lean mass (aLM; i.e., the sum of lean mass from both arms and legs): <0.789 in men, and <0.512 in women OR
   * aLM <19.75 kg in men and <15.02 kg in women
4. Willingness to be randomised to either intervention group and to follow the study protocol.

Exclusion criteria:

General

1. Unable or unwilling to provide informed consent or accept randomisation to either study group.
2. Plans to relocate out of the study area within the next 2 years or plans to be out of the study area for more than 6 consecutive weeks in the next year;
3. Residence in long-term care;
4. Household member enrolled in the study.

Clinical conditions:

1. Current diagnosis of schizophrenia, other psychotic or bipolar disorder;
2. Consumption of more than 14 alcoholic drinks per week;
3. Difficulty communicating with the study personnel due to speech, language, or (non-corrected) hearing problems;
4. Mini Mental State Examination lower than 24/30;
5. Severe osteoarthritis (e.g., awaiting joint replacement) that would interfere with the ability to participate fully in either study arm;
6. Cancer requiring treatment in the past 3 years, except for non-melanoma skin cancers or cancers that have an excellent prognosis (e.g., early stage breast or prostate cancer);
7. Lung disease requiring regular use of supplemental oxygen;
8. Inflammatory conditions requiring regular use of oral or parenteral corticosteroid agents;
9. Severe cardiovascular disease (including New York Heart Association class III or IV congestive heart failure, clinically significant valvular disease, history of cardiac arrest, presence of an implantable defibrillator, or uncontrolled angina)
10. Upper and/or lower extremity amputation;
11. Peripheral arterial disease Lériche-Fontaine 3 or 4;
12. Parkinson's disease or other progressive neurological disorder;
13. Renal disease requiring dialysis;
14. Chest pain, severe shortness of breath, or occurrence of other safety concerns during the baseline 400-metre walk test;
15. Current participation in a structured exercise programme, physical therapy or cardiopulmonary rehabilitation;
16. Current enrolment in another randomised clinical trial involving lifestyle, nutrition, or pharmaceutical interventions;
17. Other medical, psychiatric, or behavioural factors that in the judgment of the principal investigator may interfere with the study participation or the ability to autonomously follow either the multicomponent or the healthy aging lifestyle education programmes;
18. Other illness of such severity that life expectancy is expected to be less than 12 months;
19. Clinical judgment concerning safety or non-compliance.

Temporary exclusion criteria

1. Uncontrolled hypertension (systolic blood pressure >200 mm Hg, or diastolic blood pressure >110 mm Hg);
2. Uncontrolled diabetes with recent weight loss, diabetic coma, or frequent hypoglycaemia;
3. Hip fracture, hip or knee replacement, or spinal surgery in the past 6 months
4. Serious cardiac conduction disorder (e.g., third-degree heart block), uncontrolled arrhythmia, new Q waves within the past 6 months or ST-segment depression (>3 mm) on the electrocardiogram;
5. Myocardial infarction, major heart surgery (i.e., valve replacement or coronary bypass graft), stroke, deep vein thrombosis, or pulmonary embolism in the past 6 months;
6. Use of growth hormone, oestrogens, progesterone, or testosterone supplementation in the past 3 months.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Incident of major mobility disability | 36 months
  Incident inability to complete the 400-metre walk test (incidence of major mobility disability)

SECONDARY OUTCOMES:
Changes in lower extremity physical performance | 36 months
  Changes in short physical performance battery (SPPB) summary score
Changes in upper extremity muscle strength | 36 months
  Changes in handgrip strength test performance (kg)
Changes in functional status (activities of daily living) | 36 months
  Changes in Activities of Daily Living (ADL) score computed through a modified version of the Pepper Assessment Tool for Disability (PAT-D)
Changes in functional status (instrumental activities of daily living) | 36 months
  Changes in Instrumental Activities of Daily Living (IADL) score computed through a modified version of the Pepper Assessment Tool for Disability (PAT-D)
Changes in crude appendicular lean mass | 36 months
  Changes in crude in appendicular lean mass (kg) by Dual Energy X-Ray Absorptiometry
Changes in body mass index-adjusted appendicular lean mass | 36 months
  Changes in body mass index-adjusted appendicular lean mass (adimensional) by Dual Energy X-Ray Absorptiometry
Persistent mobility disability | 36 months
  Inability to complete the 400-metre walk test at two consecutive semiannual visits
Changes in body weight | 36 months
  Changes in body weight (kg)
Changes in body mass index | 36 months
  Changes in body mass index (kg/m^2)
Changes in mid-arm circumference | 36 months
  Changes in mid-arm circumference (cm)
Changes in waist circumference | 36 months
  Changes in waist circumference (cm)
Changes in hip circumference | 36 months
  Changes in hip circumference (cm)
Changes in calf circumference | 36 months
  Changes in calf circumference (cm)
Changes in nutritional status | 36 months
  Changes in Mini Nutritional Assessment-Short Form (MNA-SF) score
Changes in cognitive function | 36 months
  Changes in Mini Mental State Examination (MMSE) score
Changes in mood | 36 months
  Changes in 11-item Center for Epidemiological Studies - Depression (CES-D) scale score
Incidence of self-reported falls | 36 months
  Number of falls assessed by questionnaires
Incidence of injurious falls | 36 months
  Number of injurious falls assessed by questionnaires
Changes in quality of life | 36 months
  Changes in EuroQoL-5D (EQ5D) score
Changes in the use of healthcare services | 36 months
  Health economics questionnaire
All-cause mortality | 36 months
  Mortality rate
Cost effectiveness | 36 months
  Cost effectiveness analysis

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Landi, MD, PhD, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Catholic University of the Sacred Heart, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Coelho-Junior HJ, Alvarez-Bustos A, Rodriguez-Manas L, Landi F, Marzetti E. Comparison of muscle strength and power in the short physical performance battery for predicting negative outcomes in older adults with mobility limitations. J Nutr Health Aging. 2025 Sep;29(9):100631. doi: 10.1016/j.jnha.2025.100631. Epub 2025 Jul 15. PMID 40669418
- [Derived] Levati E, Zazzara MB, Iurlaro A, Marzetti E, Calvani R, Pahor M, Picca A, Tosato M, Landi F, Bernabei R, Onder G. Lifestyle interventions and medication burden in older adults: insights from the Lifestyle Intervention and Independence for Elders (LIFE) and the Sarcopenia and Physical fRailty iN older people: multi-componenT Treatment strategies (SPRINTT) trials. Eur Geriatr Med. 2025 Oct;16(5):1591-1598. doi: 10.1007/s41999-025-01266-0. Epub 2025 Jul 15. PMID 40665144
- [Derived] Alvarez-Bustos A, Coelho-Junior HJ, Calvani R, Rodriguez-Manas L, Tosato M, Cesari M, Cherubini A, Cruz-Jentoft AJ, Jonsson PV, Lattanzio F, Maggio M, Roller-Wirnsberger R, Ryznarova I, Schols AMWJ, Sieber CC, Sinclair AJ, Skalska A, Strandberg T, Tchalla A, Topinkova E, Vellas B, von Haehling S, Landi F, Marzetti E; SPRINTT consortium. Adherence to Physical Activity and Incident Mobility Disability in Older Adults With Mobility Limitations. J Cachexia Sarcopenia Muscle. 2025 Jun;16(3):e13870. doi: 10.1002/jcsm.13870. PMID 40532064
- [Derived] Bernabei R, Landi F, Calvani R, Cesari M, Del Signore S, Anker SD, Bejuit R, Bordes P, Cherubini A, Cruz-Jentoft AJ, Di Bari M, Friede T, Gorostiaga Ayestaran C, Goyeau H, Jonsson PV, Kashiwa M, Lattanzio F, Maggio M, Mariotti L, Miller RR, Rodriguez-Manas L, Roller-Wirnsberger R, Ryznarova I, Scholpp J, Schols AMWJ, Sieber CC, Sinclair AJ, Skalska A, Strandberg T, Tchalla A, Topinkova E, Tosato M, Vellas B, von Haehling S, Pahor M, Roubenoff R, Marzetti E; SPRINTT consortium. Multicomponent intervention to prevent mobility disability in frail older adults: randomised controlled trial (SPRINTT project). BMJ. 2022 May 11;377:e068788. doi: 10.1136/bmj-2021-068788. PMID 35545258